CLINICAL TRIAL: NCT05217641
Title: A Phase 1, Randomized, Open-label Clinical Trial to Evaluate the Safety and Immunogenicity of BG505 MD39.3, BG505 MD39.3 gp151, and BG505 MD39.3 gp151 CD4KO HIV Trimer mRNA Vaccines in Healthy, HIV-uninfected Adult Participants
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of BG505 MD39.3, BG505 MD39.3 gp151, and BG505 MD39.3 gp151 CD4KO HIV Trimer mRNA Vaccines in Healthy, HIV-uninfected Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: HVTN 302; DAIDS-ES ID: 38791 (Other: Division of AIDS)
Record Dates: First submitted 2021-12-30; First posted 2022-02-01 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: Blood-Borne Infections; Communicable Diseases; Infections; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Immunologic Factors; Physiological Effects of Drugs
MeSH Terms: conditions — HIV Infections; Blood-Borne Infections; Communicable Diseases; Infections; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Immunologic Deficiency Syndromes; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A, Group 1: Low dose BG505 MD39.3 mRNA (Experimental): 18 participants Dose: 100mcg of BG505 MD39.3 mRNA formulated administered at months 0, 2, and 6
  Interventions: Biological: BG505 MD39.3 mRNA
- Part A, Group 2: Low dose BG505 MD39.3 gp151 mRNA (Experimental): 18 participants Dose: 100mcg of BG505 MD39.3 gp151 mRNA administered at months 0, 2, and 6
  Interventions: Biological: BG505 MD39.3 gp151 mRNA
- Part A, Group 3: Low dose BG505 MD39.3 gp151 CD4KO mRNA (Experimental): 18 participants Dose: 100mcg of BG505 MD39.3 gp151 CD4KO mRNA administered at months 0, 2, and 6
  Interventions: Biological: BG505 MD39.3 gp151 CD4KO mRNA
- Part B, Group 1: BG505 MD39.3 mRNA (Experimental): 18 participants Dose: 250mcg of BG505 MD39.3 mRNA administered at months 0, 2, and 6
  Interventions: Biological: BG505 MD39.3 mRNA
- Part B, Group 2: BG505 MD39.3 gp151 mRNA (Experimental): 18 participants Dose: 250mcg of BG505 MD39.3 gp151 mRNA administered at months 0, 2, and 6
  Interventions: Biological: BG505 MD39.3 gp151 mRNA
- Part B, Group 3: BG505 MD39.3 gp151 CD4KO mRNA (Experimental): 18 participants Dose: 250mcg of BG505 MD39.3 gp151 CD4KO mRNA administered at months 0, 2, and 6
  Interventions: Biological: BG505 MD39.3 gp151 CD4KO mRNA

INTERVENTIONS:
Biological: BG505 MD39.3 mRNA — Administered by IM injection
  Arms: Part A, Group 1: Low dose BG505 MD39.3 mRNA; Part B, Group 1: BG505 MD39.3 mRNA
Biological: BG505 MD39.3 gp151 mRNA — Administered by IM injection
  Arms: Part A, Group 2: Low dose BG505 MD39.3 gp151 mRNA; Part B, Group 2: BG505 MD39.3 gp151 mRNA
Biological: BG505 MD39.3 gp151 CD4KO mRNA — Administered by IM injection
  Arms: Part A, Group 3: Low dose BG505 MD39.3 gp151 CD4KO mRNA; Part B, Group 3: BG505 MD39.3 gp151 CD4KO mRNA

SUMMARY:
This is an open-label, multicenter, randomized phase 1 study to evaluate the safety and immunogenicity of BG505 MD39.3, BG505 MD39.3 gp151, and BG505 MD39.3 gp151 CD4KO HIV trimer mRNA. These trimers are based on the BG505 MD39 native-like trimer reported in Steichen et al. Immunity 2016. The primary hypothesis is that the BG505 MD39.3 soluble and membrane-bound trimer mRNA vaccines will be safe and well-tolerated among HIV-uninfected individuals and will elicit autologous neutralizing antibodies.

DETAILED DESCRIPTION:
Participants will receive BG505 MD39.3 mRNA, BG505 MD39.3 gp151 mRNA or BG505 MD39.3 gp151 CD4KO mRNA, at doses of 100 mcg or 250mcg, administered via intramuscular (IM) injections into the deltoid muscle. Participants will be evaluated for safety and immune responses through blood and lymph node fine-needle aspiration collection at specified timepoints throughout the study.

A dose escalation plan will be implemented, whereby sentinel safety groups for each of the three low-dose groups in Part A would be enrolled and evaluated for safety 2 weeks after the first vaccination. If safety criteria are met, then enrollment of the Part B sentinel safety groups and the remainder of the Part A participants would commence. Safety for the sentinel groups in Part B will be assessed after the first vaccination prior to full enrollment of Part B. In addition, standard safety evaluations will occur routinely throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete the informed consent process, including an Assessment of Understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly.
2. 18-55 years old, inclusive, on day of enrollment.
3. Agrees to comply with planned study procedures and be available for clinic follow-up through the last clinic visit.
4. Agrees not to enroll in another study of an investigational agent during participation in the trial.
5. In good general health according to the clinical judgement of the site investigator.
6. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
7. Assessed as low risk for HIV acquisition per low risk guidelines, agrees to discuss HIV infection risks, agrees to risk reduction counseling, and agrees to avoid behavior associated with high risk of HIV exposure through the final study visit. Low risk may include persons stably taking pre-exposure prophylaxis (PrEP) as prescribed for 6 months or longer.
8. Hemoglobin

   * Greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth
   * Greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth and transgender males who have been on hormone therapy for more than 6 consecutive months
   * Greater than or equal to 12.0 g/dL for transgender females who have been on hormone therapy for more than 6 consecutive months
   * For transgender participants who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth
9. White blood cell (WBC) count > 3,500/mm3
10. Platelets ≥125,000 /mm3
11. Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) based on the institutional normal range
12. Serum creatinine ≤1.1 x ULN based on the institutional normal range
13. Negative results for HIV infection by an (US) Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
14. Negative for anti-Hepatitis C antibodies (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies are detected.
15. Negative for Hepatitis B surface antigen.
16. For a volunteer capable of becoming pregnant:

    * Volunteers who were assigned female sex at birth and are of reproductive potential must agree to use effective means of birth control from at least 21 days prior to enrollment through 3 months after their third vaccination timepoint
    * Has negative β-HCG (beta human chorionic gonadotropin) pregnancy test (urine or serum) at screening and prior to study product administration on day of enrollment.

Exclusion Criteria:

1. Volunteer who is breast-feeding or pregnant.
2. Hypertension that is not well controlled. If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently < 140 mm Hg systolic and < 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be < 140 mm Hg systolic and < 90 mm Hg diastolic at enrollment. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
3. Diabetes mellitus type 1 or type 2. (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes).
4. Previous or current recipient of an investigational HIV vaccine (previous placebo recipients are not excluded).
5. Acutely ill or febrile (temperature ≥ 38.0°C/100.4°F) on the day of the first vaccination. Participants meeting this criterion may be rescheduled within the enrollment window period. Afebrile participants with minor illnesses can be enrolled at the discretion of the Investigator.
6. Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment).
7. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
8. Receipt of any of the following:

   * Within 4 weeks prior to enrollment:

     * Any licensed live, attenuated vaccine
     * Any emergency use authorized (EUA) or licensed mRNA-based SARS-CoV-2 vaccine
   * Within 2 weeks prior to enrollment:

     * Any licensed killed/subunit/inactivated vaccine
     * Any EUA or licensed adenoviral-vectored or protein SARS-CoV-2 vaccines Receipt of any SARS-CoV-2 vaccination series should be completed 4 weeks prior to enrollment when possible; however, exceptions may be made by approval of the HVTN 302 PSRT.
9. Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
10. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
11. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any vaccine or any component of the study vaccine.
12. History of myocarditis and/or pericarditis.
13. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
14. Idiopathic urticaria within the past year.
15. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
16. Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
17. Asplenia or functional asplenia.
18. Active duty and reserve US military personnel.
19. Any other chronic or clinically significant condition that in the clinical judgement of the investigator would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of drug or alcohol abuse, serious psychiatric disorders, or cancer that, in the clinical judgement of the site investigator, has a potential for recurrence (excluding basal cell carcinoma).
20. Asthma is excluded if the participant has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or co-existing conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
    * Uses more than one medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than one medication for maintenance therapy daily for greater than two years requires PSRT approval.
21. A participant with a history of an immune-mediated disease, either active or remote. Not exclusionary: 1) remote history of Bell's palsy (>2 years ago) not associated with other neurologic symptoms, 2) mild psoriasis that does not require ongoing systemic treatment.
22. Immunodeficiency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2027-06-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Clark, MD, Study Chair — University of California, Los Angeles; Sharon Riddler, MD, Study Chair — University of Pittsburgh
Locations (10):
- United States (10):
  - Alabama CRS [31788], Birmingham, Alabama
  - UCLA Vine Street Clinic CRS [31607], Los Angeles, California
  - Bidmc Vcrs [32077], Boston, Massachusetts
  - Brigham and Women's Hospital Vaccine CRS [30007], Boston, Massachusetts
  - New York Blood Center CRS [31801], New York, New York
  - Columbia P&S CRS [30329], New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS [31467], Rochester, New York
  - Penn Prevention CRS [30310], Philadelphia, Pennsylvania
  - University of Pittsburgh CRS [1001], Pittsburgh, Pennsylvania
  - Seattle Vaccine and Prevention CRS [30331], Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riddler SA, Moodie Z, Clark J, Yen C, Allen M, Furch BD, Lu H, Grant S, Mondal K, Anderson M, Maenza J, Lemos MP, Woodward Davis AS, Walsh SR, Sobieszczyk ME, Frank I, Goepfert P, Stephenson KE, Baden LR, Tieu HV, Keefer MC, McElrath MJ, Kublin JG, Corey L. High Frequency of Chronic Urticaria Following an Investigational HIV-1 BG505 MD39.3 Trimer mRNA Vaccine in a Phase 1, Randomized, Open-Label Clinical Trial (HVTN 302). Ann Intern Med. 2025 Jul;178(7):963-974. doi: 10.7326/ANNALS-24-02701. Epub 2025 Apr 29. PMID 40294415

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Group 1: Treatment: 100 mcg of BG505 MD39.3 mRNA
- Part A, Group 2: Treatment: 100 mcg of BG505 MD39.3 gp151 mRNA
- Part A, Group 3: Treatment: 100 mcg of BG505 MD39.3 gp151 CD4KO mRNA
- Part B, Group 4: Treatment: 250 mcg of BG505 MD39.3 mRNA
- Part B, Group 5: Treatment: 250 mcg of BG505 MD39.3 gp151 mRNA
- Part B, Group 6: Treatment: 250 mcg of BG505 MD39.3 gp151 CD4KO mRNA
Period: Overall Study
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Started | 18 | 19 | 17 | 18 | 18 | 18
Completed | 16 | 17 | 17 | 14 | 14 | 18
Not Completed | 2 | 2 | 0 | 4 | 4 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Other: participant did not specify reason | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Extended Follow up | 1 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment | Total
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18 | 108
Age, Continuous [Median (Full Range); unit: years] | 25.5 [19 to 41] | 35 [19 to 54] | 31 [18 to 55] | 27 [19 to 42] | 26 [18 to 49] | 30 [20 to 48] | 28.5 [18 to 55]
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 years | 3 | 2 | 1 | 1 | 2 | 3 | 12
  21 - 30 years | 10 | 4 | 7 | 12 | 11 | 7 | 51
  31 - 40 years | 4 | 10 | 6 | 4 | 3 | 5 | 32
  41 - 50 years | 1 | 1 | 2 | 1 | 2 | 3 | 10
  Over 50 years | 0 | 2 | 1 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 7 | 9 | 7 | 7 | 52
  Male | 6 | 9 | 10 | 9 | 11 | 11 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 1 | 2 | 3 | 3 | 18
  Not Hispanic or Latino | 10 | 18 | 16 | 16 | 15 | 15 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 2 | 2 | 0 | 2 | 15
  White | 14 | 12 | 13 | 12 | 18 | 15 | 84
  More than one race | 1 | 0 | 1 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  US | 18 | 19 | 17 | 18 | 18 | 18 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, July 2017. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 7 days after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  None | 0 | 1 | 1 | 0 | 0 | 0
  Mild | 10 | 7 | 9 | 8 | 8 | 10
  Moderate | 8 | 10 | 4 | 8 | 9 | 8
  Severe | 0 | 1 | 3 | 2 | 1 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Unsolicited Adverse Events Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 7 days after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  Erythema/Redness: None | 17 | 13 | 16 | 16 | 15 | 12
  Erythema/Redness: Mild | 1 | 1 | 0 | 1 | 1 | 2
  Erythema/Redness: Moderate | 0 | 4 | 1 | 0 | 2 | 3
  Erythema/Redness: Severe | 0 | 1 | 0 | 1 | 0 | 1
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 16 | 15 | 12 | 14 | 17 | 14
  Induration/Swelling: Mild | 0 | 1 | 2 | 1 | 1 | 1
  Induration/Swelling: Moderate | 2 | 3 | 2 | 2 | 0 | 3
  Induration/Swelling: Severe | 0 | 0 | 1 | 1 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 15 | 13 | 12 | 13 | 14 | 12
  Erythema and/or Induration: Mild | 1 | 1 | 2 | 2 | 2 | 1
  Erythema and/or Induration: Moderate | 2 | 4 | 2 | 2 | 2 | 4
  Erythema and/or Induration: Severe | 0 | 1 | 1 | 1 | 0 | 1
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through 7 days after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  Malaise and/or fatigue: None | 2 | 7 | 2 | 3 | 0 | 3
  Malaise and/or fatigue: Mild | 11 | 6 | 7 | 6 | 8 | 1
  Malaise and/or fatigue: Moderate | 5 | 2 | 6 | 7 | 8 | 12
  Malaise and/or fatigue: Severe | 0 | 4 | 2 | 2 | 2 | 2
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 5 | 11 | 5 | 7 | 0 | 0
  Myalgia: Mild | 8 | 3 | 7 | 3 | 10 | 8
  Myalgia: Moderate | 5 | 3 | 3 | 6 | 8 | 10
  Myalgia: Severe | 0 | 2 | 2 | 2 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 4 | 6 | 3 | 3 | 1 | 1
  Headache: Mild | 11 | 8 | 10 | 11 | 10 | 9
  Headache: Moderate | 3 | 3 | 2 | 4 | 5 | 7
  Headache: Severe | 0 | 2 | 2 | 0 | 2 | 1
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 14 | 16 | 9 | 11 | 9 | 8
  Nausea: Mild | 4 | 1 | 5 | 6 | 6 | 6
  Nausea: Moderate | 0 | 2 | 3 | 1 | 3 | 4
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 7 | 13 | 6 | 11 | 2 | 5
  Chills: Mild | 8 | 2 | 8 | 5 | 9 | 6
  Chills: Moderate | 3 | 1 | 2 | 2 | 7 | 7
  Chills: Severe | 0 | 3 | 1 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 10 | 10 | 5 | 11 | 8 | 7
  Arthralgia: Mild | 6 | 7 | 7 | 7 | 5 | 7
  Arthralgia: Moderate | 2 | 1 | 4 | 0 | 4 | 4
  Arthralgia: Severe | 0 | 1 | 1 | 0 | 1 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 1 | 4 | 1 | 0 | 0 | 0
  Max. Systemic Symptoms: Mild | 10 | 9 | 7 | 8 | 3 | 3
  Max. Systemic Symptoms: Moderate | 7 | 1 | 6 | 7 | 11 | 13
  Max. Systemic Symptoms: Severe | 0 | 5 | 3 | 3 | 4 | 2
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 14 | 13 | 17 | 17 | 12 | 9
  Temperature: Mild | 4 | 5 | 0 | 0 | 4 | 7
  Temperature: Moderate | 0 | 0 | 0 | 0 | 2 | 2
  Temperature: Severe | 0 | 1 | 0 | 1 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - ALT in U/L
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population
Time Frame: Measured during Screening, Days 8, 64, 176 and 225
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
U/L
  ALT (U/L) -Screening | 15 [13 to 21] | 17 [12 to 23] | 17 [15 to 28] | 15 [12 to 25] | 19 [13 to 23] | 23 [17 to 31]
  ALT (U/L) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  ALT (U/L) -V3 - 1 week post-vaccination 1 | 14 [11 to 19] | 16 [14 to 25] | 17 [13 to 32] | 14.5 [14 to 30] | 14.5 [12 to 20] | 20 [17 to 24]
  ALT (U/L) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  ALT (U/L) -V7 - 1 week post-vaccination 2 | 13 [12 to 16] | 17 [13 to 22.5] | 17 [12 to 31] | 14 [12 to 19] | 15 [11 to 19] | 22 [17.5 to 35.5]
  ALT (U/L) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  ALT (U/L) -V11 - 1 week post-Vaccination 3 | 12 [11 to 18] | 13 [10 to 19] | 13 [12 to 29] | 12 [10 to 17] | 13 [12 to 17] | 19 [15 to 24]
  ALT (U/L) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  ALT (U/L) -V14 - 8 weeks post-vaccination 3 |  |  |  | 28 [28 to 28] |  |

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine in mg/dL
Description: as for outcome 4
Time Frame: Measured during Screening, Days 8, 64, 176 and 225
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
mg/dL
  Creatinine (mg/dL) -Screening | 0.82 [0.66 to 0.89] | 0.91 [0.79 to 1.05] | 0.87 [0.8 to 0.91] | 0.79 [0.68 to 0.91] | 0.91 [0.76 to 0.98] | 0.86 [0.73 to 0.94]
  Creatinine (mg/dL) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Creatinine (mg/dL) -V3 - 1 week post-vaccination 1 | 0.77 [0.67 to 0.86] | 0.9 [0.79 to 1.1] | 0.91 [0.79 to 0.98] | 0.76 [0.71 to 0.96] | 0.91 [0.79 to 1] | 0.82 [0.74 to 1.03]
  Creatinine (mg/dL) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Creatinine (mg/dL) -V7 - 1 week post-vaccination 2 | 0.8 [0.71 to 0.86] | 1 [0.86 to 1.09] | 0.84 [0.8 to 0.93] | 0.76 [0.68 to 0.88] | 0.9 [0.82 to 0.96] | 0.87 [0.76 to 0.95]
  Creatinine (mg/dL) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Creatinine (mg/dL) -V11 - 1 week post-Vaccination 3 | 0.83 [0.71 to 0.91] | 0.95 [0.8 to 1.09] | 0.86 [0.75 to 1] | 0.8 [0.62 to 0.88] | 0.86 [0.77 to 0.92] | 0.81 [0.74 to 1.03]
  Creatinine (mg/dL) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine (mg/dL) -V14 - 8 weeks post-vaccination 3 |  |  |  | 0.83 [0.83 to 0.83] |  |

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin in g/dL
Description: as for outcome 4
Time Frame: Measured during Screening, Days 8, 64, 176 and 225
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
g/dL
  Hemoglobin (g/dL) -Screening | 14.55 [12.9 to 15.1] | 13.7 [12.9 to 15.6] | 14.2 [12.9 to 14.9] | 14.1 [13.4 to 15] | 14.75 [14.1 to 15.7] | 14.15 [13.2 to 15]
  Hemoglobin (g/dL) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Hemoglobin (g/dL) -V3 - 1 week post-vaccination 1 | 13.8 [12.9 to 14.4] | 13.8 [12.9 to 15.4] | 13.7 [12.7 to 14.5] | 13.85 [13 to 15.2] | 14.1 [13.8 to 15.1] | 13.8 [13.1 to 14.9]
  Hemoglobin (g/dL) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Hemoglobin (g/dL) -V7 - 1 week post-vaccination 2 | 13.5 [11.8 to 14.6] | 13.65 [12.6 to 14.85] | 13.4 [12.2 to 14.4] | 13.1 [12.6 to 13.8] | 13.8 [13.1 to 14.5] | 14 [12.45 to 15]
  Hemoglobin (g/dL) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Hemoglobin (g/dL) -V11 - 1 week post-Vaccination 3 | 13.7 [11.9 to 14.4] | 13.5 [12 to 14.5] | 13.7 [12.3 to 14.2] | 12.9 [12.4 to 13.3] | 13.7 [12.9 to 14.5] | 13.2 [12.4 to 14.5]
  Hemoglobin (g/dL) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Hemoglobin (g/dL) -V14 - 8 weeks post-vaccination 3 | 13.7 [12.2 to 14.3] | 13.4 [11.7 to 14.3] | 13.9 [12.3 to 14.6] | 12.9 [11.7 to 13.5] | 13.7 [12.2 to 14.8] | 13.25 [12.65 to 14.5]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil, Basophils, Eosinophils Count in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during Screening, Days 8, 64, 176 and 225
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/Cubic mm
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
1000 cells/Cubic mm
  Lymphocytes (1000 cells/Cubic mm) -Screening | 2.12 [1.78 to 2.36] | 1.93 [1.8 to 2.68] | 1.86 [1.55 to 2.1] | 2.05 [1.46 to 2.6] | 1.79 [1.56 to 2.18] | 1.78 [1.31 to 2.25]
  Lymphocytes (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Lymphocytes (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1 | 2.02 [1.74 to 2.3] | 1.92 [1.6 to 2.57] | 1.85 [1.66 to 2.37] | 2.08 [1.65 to 2.48] | 1.9 [1.47 to 2.2] | 1.89 [1.64 to 2.09]
  Lymphocytes (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Lymphocytes (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2 | 2.17 [1.68 to 2.5] | 2.08 [1.83 to 2.27] | 1.85 [1.62 to 2.19] | 2.1 [1.57 to 2.32] | 1.9 [1.66 to 2.45] | 1.87 [1.54 to 2.22]
  Lymphocytes (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Lymphocytes (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3 | 2.02 [1.69 to 2.51] | 2.1 [1.69 to 2.53] | 1.85 [1.6 to 2.24] | 2.01 [1.92 to 2.2] | 2.02 [1.69 to 2.31] | 2.04 [1.81 to 2.21]
  Lymphocytes (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Lymphocytes (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3 | 1.79 [1.49 to 2.03] | 1.86 [1.56 to 2.14] | 1.78 [1.59 to 2.21] | 1.94 [1.69 to 2.18] | 2.13 [1.66 to 2.23] | 1.95 [1.73 to 2.16]
  Neutrophils (1000 cells/Cubic mm) -Screening | 4.26 [2.97 to 4.81] | 3.39 [2.66 to 4.28] | 3.9 [3.54 to 5.73] | 4.13 [3.42 to 5.4] | 3.31 [2.56 to 4.35] | 3.22 [2.31 to 5]
  Neutrophils (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Neutrophils (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1 | 3.9 [2.81 to 4.65] | 3.84 [2.77 to 5.14] | 3.53 [2.91 to 4.93] | 3.33 [2.45 to 4.9] | 3.44 [2.88 to 4.21] | 3.59 [2.66 to 4.3]
  Neutrophils (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Neutrophils (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2 | 3.54 [3.02 to 4.4] | 3.07 [2.8 to 4.05] | 3.07 [2.52 to 3.9] | 3.37 [2.66 to 4.24] | 2.73 [2.21 to 3.56] | 2.86 [2.25 to 4.38]
  Neutrophils (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Neutrophils (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3 | 3.09 [2.43 to 4.76] | 3.18 [2.34 to 4.65] | 3.67 [2.4 to 4.89] | 3.2 [2.4 to 3.79] | 2.8 [1.99 to 3.38] | 3.18 [2.89 to 3.64]
  Neutrophils (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Neutrophils (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3 | 3.5 [3.29 to 4.91] | 3.76 [3.37 to 5.65] | 3.6 [2.93 to 5.31] | 3.01 [2.62 to 3.79] | 2.73 [2.11 to 4.77] | 3.42 [3.22 to 4.71]
  Basophils (1000 cells/Cubic mm) -Screening | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.07] | 0.05 [0.03 to 0.05] | 0.05 [0.04 to 0.07] | 0.04 [0.03 to 0.07] | 0.04 [0.03 to 0.06]
  Basophils (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Basophils (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1 | 0.04 [0.04 to 0.06] | 0.05 [0.03 to 0.07] | 0.05 [0.04 to 0.07] | 0.05 [0.03 to 0.06] | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05]
  Basophils (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Basophils (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2 | 0.04 [0.03 to 0.06] | 0.05 [0.04 to 0.06] | 0.05 [0.03 to 0.06] | 0.04 [0.02 to 0.05] | 0.05 [0.03 to 0.07] | 0.04 [0.03 to 0.05]
  Basophils (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Basophils (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3 | 0.05 [0.04 to 0.06] | 0.06 [0.04 to 0.06] | 0.05 [0.04 to 0.07] | 0.05 [0.03 to 0.06] | 0.05 [0.03 to 0.07] | 0.04 [0.03 to 0.06]
  Basophils (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Basophils (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3 | 0.04 [0.03 to 0.05] | 0.05 [0.04 to 0.07] | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05] | 0.05 [0.02 to 0.07] | 0.03 [0.02 to 0.05]
  Eosinophils (1000 cells/Cubic mm) -Screening | 0.08 [0.05 to 0.1] | 0.11 [0.09 to 0.17] | 0.12 [0.06 to 0.16] | 0.11 [0.07 to 0.2] | 0.14 [0.1 to 0.22] | 0.12 [0.09 to 0.17]
  Eosinophils (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Eosinophils (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1 | 0.16 [0.1 to 0.25] | 0.12 [0.1 to 0.17] | 0.18 [0.1 to 0.3] | 0.16 [0.12 to 0.28] | 0.21 [0.14 to 0.3] | 0.19 [0.1 to 0.3]
  Eosinophils (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Eosinophils (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2 | 0.14 [0.07 to 0.21] | 0.13 [0.1 to 0.22] | 0.15 [0.11 to 0.25] | 0.17 [0.13 to 0.3] | 0.2 [0.15 to 0.26] | 0.19 [0.11 to 0.25]
  Eosinophils (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Eosinophils (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3 | 0.11 [0.09 to 0.18] | 0.15 [0.11 to 0.18] | 0.13 [0.1 to 0.2] | 0.11 [0.1 to 0.26] | 0.2 [0.17 to 0.38] | 0.14 [0.1 to 0.21]
  Eosinophils (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Eosinophils (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3 | 0.1 [0.07 to 0.13] | 0.11 [0.07 to 0.17] | 0.13 [0.11 to 0.19] | 0.13 [0.07 to 0.22] | 0.18 [0.12 to 0.26] | 0.11 [0.08 to 0.15]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during Screening, Days 8, 64, 176 and 225
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/Cubic mm
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
1000 cells/Cubic mm
  WBC (1000 cells/Cubic mm) -Screening | 7.05 [5.46 to 7.78] | 6.23 [5.41 to 6.47] | 6.76 [6.08 to 8.17] | 7.1 [6 to 8.5] | 5.82 [4.91 to 7.5] | 6.25 [4.3 to 8.36]
  WBC (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  WBC (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1 | 6.45 [5.63 to 7.86] | 6.7 [5.1 to 7.7] | 6.7 [5.6 to 8.36] | 6.17 [5.4 to 7.36] | 6.09 [5 to 7.1] | 6.14 [5.1 to 7.22]
  WBC (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  WBC (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2 | 6.17 [5.5 to 8.33] | 5.79 [5.15 to 7.2] | 5.65 [5.19 to 6.22] | 6.64 [5.1 to 7] | 5.7 [4.44 to 6.8] | 5.43 [4.54 to 7.3]
  WBC (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  WBC (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3 | 5.59 [4.95 to 7.42] | 6.21 [5.25 to 7.12] | 6.64 [5.1 to 7.69] | 6 [5.1 to 6.7] | 5.49 [4.3 to 6.3] | 5.9 [5.7 to 7.6]
  WBC (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  WBC (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3 | 5.99 [5.6 to 7.3] | 6.49 [5.08 to 7.8] | 6.1 [5.12 to 7.84] | 5.91 [4.96 to 6.6] | 5.71 [4.75 to 8.53] | 6.26 [5.65 to 7.42]
  Platelets (1000 cells/Cubic mm) -Screening | 257 [223 to 282] | 267 [249 to 330] | 284 [237 to 325] | 276 [261 to 299] | 257.5 [208 to 308] | 259 [222 to 305]
  Platelets (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Platelets (1000 cells/Cubic mm) -V3 - 1 week post-vaccination 1 | 251 [216 to 306] | 277 [254 to 342] | 287 [236 to 331] | 283.5 [244 to 316] | 256.5 [217 to 321] | 281 [240 to 292]
  Platelets (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Platelets (1000 cells/Cubic mm) -V7 - 1 week post-vaccination 2 | 271 [244 to 305] | 285.5 [238.5 to 349] | 267 [232 to 306] | 279 [264 to 288] | 262 [237 to 352] | 278 [240 to 309.5]
  Platelets (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Platelets (1000 cells/Cubic mm) -V11 - 1 week post-Vaccination 3 | 267.3 [228.5 to 294] | 269 [250 to 341] | 275 [256 to 326] | 295 [267 to 319] | 271 [239 to 367] | 274 [249 to 312]
  Platelets (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Platelets (1000 cells/Cubic mm) -V14 - 8 weeks post-vaccination 3 | 290 [232 to 327] | 277 [242 to 325.3] | 279 [255 to 314] | 271.5 [247 to 315] | 291 [214 to 351] | 281 [249 to 316]

9. Primary Outcome: Number of Lab Grade > 1 for ALT, Creatinine, Hemoglobin, Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC), Basophils, Eosinophils
Description: The number (percentage) of participants with lab grade > 1 for alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC), basophils, eosinophils was summarized by arm
Time Frame: Measured during Screening, Days 8, 64, 176 and 225
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  ALT (U/L) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  ALT (U/L) -V3 - 1 week post-vaccination 1 | 1 | 0 | 0 | 1 | 1 | 1
  ALT (U/L) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  ALT (U/L) -V7 - 1 week post-vaccination 2 | 1 | 0 | 0 | 1 | 1 | 0
  ALT (U/L) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  ALT (U/L) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 1 | 0 | 0
  ALT (U/L) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  ALT (U/L) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Hemoglobin (g/dL) -V3 - 1 week post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Hemoglobin (g/dL) -V7 - 1 week post-vaccination 2 | 0 | 0 | 2 | 0 | 0 | 1
  Hemoglobin (g/dL) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Hemoglobin (g/dL) -V11 - 1 week post-Vaccination 3 | 0 | 1 | 1 | 0 | 0 | 0
  Hemoglobin (g/dL) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Hemoglobin (g/dL) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 2 | 0 | 0 | 0
  Creatinine (mg/dL) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Creatinine (mg/dL) -V3 - 1 week post-vaccination 1 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Creatinine (mg/dL) -V7 - 1 week post-vaccination 2 | 0 | 1 | 0 | 0 | 0 | 1
  Creatinine (mg/dL) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Creatinine (mg/dL) -V11 - 1 week post-Vaccination 3 | 0 | 1 | 1 | 1 | 0 | 0
  Creatinine (mg/dL) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine (mg/dL) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  WBC (1000/cubic mm) -V3 - 1 week post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  WBC (1000/cubic mm) -V7 - 1 week post-vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  WBC (1000/cubic mm) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  WBC (1000/cubic mm) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Platelets (1000/cubic mm) -V3 - 1 week post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Platelets (1000/cubic mm) -V7 - 1 week post-vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Platelets (1000/cubic mm) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Platelets (1000/cubic mm) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Lymphocytes (1000/cubic mm) -V3 - 1 week post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Lymphocytes (1000/cubic mm) -V7 - 1 week post-vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Lymphocytes (1000/cubic mm) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Lymphocytes (1000/cubic mm) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Neutrophils (1000/cubic mm) -V3 - 1 week post-vaccination 1 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Neutrophils (1000/cubic mm) -V7 - 1 week post-vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Neutrophils (1000/cubic mm) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Neutrophils (1000/cubic mm) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (1000/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (1000/cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Basophils (1000/cubic mm) -V3 - 1 week post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (1000/cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Basophils (1000/cubic mm) -V7 - 1 week post-vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (1000/cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Basophils (1000/cubic mm) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils (1000/cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Basophils (1000/cubic mm) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (1000/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (1000/cubic mm) -V3 - 1 week post-vaccination 1: number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 17
  Eosinophils (1000/cubic mm) -V3 - 1 week post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (1000/cubic mm) -V7 - 1 week post-vaccination 2: number analyzed (Participants) | 17 | 16 | 16 | 13 | 17 | 16
  Eosinophils (1000/cubic mm) -V7 - 1 week post-vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (1000/cubic mm) -V11 - 1 week post-Vaccination 3: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 17
  Eosinophils (1000/cubic mm) -V11 - 1 week post-Vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (1000/cubic mm) -V14 - 8 weeks post-vaccination 3: number analyzed (Participants) | 17 | 17 | 17 | 14 | 15 | 16
  Eosinophils (1000/cubic mm) -V14 - 8 weeks post-vaccination 3 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Time Frame: 30 days following each injection
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  Mild | 6 | 3 | 3 | 6 | 3 | 8
  Moderate | 10 | 9 | 9 | 9 | 5 | 5
  Severe | 0 | 2 | 1 | 0 | 0 | 1
  Potentially life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0
  No AE reported | 2 | 5 | 4 | 3 | 10 | 4

11. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: as for outcome 10
Time Frame: 30 days following each injection
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  Related | 8 | 2 | 2 | 3 | 3 | 4
  Not Related | 8 | 12 | 11 | 12 | 5 | 10
  No AE reported | 2 | 5 | 4 | 3 | 10 | 4

12. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: as for outcome 10
Time Frame: Measured through Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants | 1 | 1 | 1 | 0 | 0 | 0

13. Primary Outcome: Number of Participants Reporting Medically Attended Adverse Events (MAAEs)
Description: as for outcome 10
Time Frame: Measured through Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants | 9 | 9 | 8 | 6 | 5 | 3

14. Primary Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs)
Description: There were no adverse events of special interest reported by any participant.
Time Frame: Measured through Month 12.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: as for outcome 10
Time Frame: Measured through Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  Adverse event | 2 | 1 | 0 | 1 | 1 | 1
  Reactogenicity symptom | 0 | 0 | 0 | 1 | 0 | 0
  Other reason | 0 | 2 | 0 | 7 | 3 | 1
  No Discontinuation | 16 | 16 | 17 | 9 | 14 | 16

16. Primary Outcome: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: There were no early study terminations associated with an AE or reactogenicity reported by any participant.
Time Frame: Measured through Month 12.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Magnitude of Serum Antibody Neutralization of a Vaccine-matched Tier 2 HIV-1 Strain
Description: Neutralizing antibodies against HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl cells. The assay performed in TZM-bl cells measured neutralization titers against a panel of autologous Env-pseudotyped viruses that exhibit tier 2 neutralization phenotype: BG505/T332N.
Time Frame: 2 weeks after the 3rd vaccination timepoint (M6.5)
Population: In this report, the overall number of participants analyzed represents the enrolled participants at 2 weeks after the 3rd vaccination. The Number Analyzed in the Outcome Measure Data Table shows the number of participants with available NAb data after filtering for assay specific quality control criteria.
Measure: Median (Inter-Quartile Range); unit: log10(titer)
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
log10(titer)
  BG505/T332N, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 14 | 17
  BG505/T332N, 1: 50, M6.5 | 5 [5 to 5] | 15.5 [5 to 43.6] | 35.4 [9.1 to 115.7] | 5 [5 to 5] | 73.4 [22.3 to 218.9] | 68.6 [53.2 to 348.4]
  BG505/T332N, 1: 80, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 14 | 17
  BG505/T332N, 1: 80, M6.5 | 5 [5 to 5] | 5 [5 to 13.7] | 9.6 [5 to 30.9] | 5 [5 to 5] | 22.5 [7 to 69.4] | 24.8 [15.9 to 143.3]

18. Primary Outcome: Response Rate of Serum Antibody Neutralization of a Vaccine-matched Tier 2 HIV-1 Strain
Description: as for outcome 17
Time Frame: 2 weeks after the 3rd vaccination timepoint (M6.5)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  BG505/T332N, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 14 | 17
  BG505/T332N, 1: 50, M6.5 | 0 | 11 | 12 | 1 | 12 | 16
  BG505/T332N, 1: 80, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 14 | 17
  BG505/T332N, 1: 80, M6.5 | 0 | 7 | 8 | 0 | 10 | 14

19. Secondary Outcome: Magnitude of Serum Antibody Neutralization of a Vaccine-matched Tier 2 HIV-1 Strain
Description: as for outcome 17
Time Frame: 2 weeks after the 2nd vaccination (M2.5), 6 months after the 3rd vaccination (M12)
Population: In this report, the overall number of participants analyzed represents the enrolled participants at 2 weeks after the 2nd vaccination and 6 months after the 3rd vaccination. The Number Analyzed in the Outcome Measure Data Table shows the number of participants with available NAb data after filtering for assay specific quality control criteria.
Measure: Median (Inter-Quartile Range); unit: log10(titer)
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
log10(titer)
  BG505/T332N, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 12 | 17 | 18
  BG505/T332N, 1: 50, M2.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 23.8] | 5 [5 to 5] | 5 [5 to 13.1] | 5 [5 to 5]
  BG505/T332N, 1: 50, M12: number analyzed (Participants) | 0 | 4 | 6 | 0 | 8 | 9
  BG505/T332N, 1: 50, M12 |  | 27.6 [20.7 to 47.9] | 49 [43.3 to 69.7] |  | 76.4 [36.5 to 167.2] | 67.5 [37.6 to 334.7]
  BG505/T332N, 1: 80, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 12 | 17 | 18
  BG505/T332N, 1: 80, M2.5 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  BG505/T332N, 1: 80, M12: number analyzed (Participants) | 0 | 4 | 6 | 0 | 8 | 9
  BG505/T332N, 1: 80, M12 |  | 5 [5 to 12] | 12.7 [6.6 to 18.3] |  | 22.1 [11.2 to 22.9] | 16.8 [13.8 to 57.3]

20. Secondary Outcome: Response Rate of Serum Antibody Neutralization of a Vaccine-matched Tier 2 HIV-1 Strain
Description: Neutralizing antibodies against HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl cells. The assay performed in TZM-bl cells measured neutralization titers against a panel of autologous and Env-pseudotyped viruses that exhibit tier 2 neutralization phenotype: BG505/T332N.
Time Frame: 2 weeks after the 2nd vaccination (M2.5), 6 months after the 3rd vaccination (M12)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  BG505/T332N, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 12 | 17 | 18
  BG505/T332N, 1: 50, M2.5 | 0 | 2 | 5 | 0 | 5 | 4
  BG505/T332N, 1: 50, M12: number analyzed (Participants) | 0 | 4 | 6 | 0 | 8 | 9
  BG505/T332N, 1: 50, M12 | 0 | 3 | 6 | 0 | 8 | 9
  BG505/T332N, 1: 80, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 12 | 17 | 18
  BG505/T332N, 1: 80, M2.5 | 0 | 0 | 3 | 0 | 1 | 1
  BG505/T332N, 1: 80, M12: number analyzed (Participants) | 0 | 4 | 6 | 0 | 8 | 9
  BG505/T332N, 1: 80, M12 | 0 | 1 | 4 | 0 | 6 | 7

21. Secondary Outcome: Magnitude of Serum IgG Binding Antibodies to the BG505 Trimer, and Specific Epitopes (Base of Trimer, V3, Internal Epitope) as Measured by Binding Antibody Multiplex Assay (BAMA)
Description: Serum HIV-1 specific IgG responses against BG505 MD39.3 trimer and BG505 MD39.3 CD4KO trimer were measured on a BioPlex instrument using a standardized custom HIV-1 Luminex assay. The readout was background subtracted mean fluorescence intensity (MFI), where background referred to a plate level control. Serum samples from post enrollment visits were declared to have positive direct binding responses if they met three conditions: 1) MFI* ≥antigen specific positivity threshold (based on the 95th percentile of baseline samples and at least 100 MFI*), 2) MFI* > 3x(Visit 2 MFI* ), and 3) MFI > 3x(Visit 2 MFI). MFI = Mean Fluorescent Intensity minus a plate specific background measure, MFI* = MFI Blank, where 'Blank' is a sample specific background measure. Results from samples with high sample background (Blank>5000 MFI), high baseline (Baseline>6500 MFI*) are excluded. MFI* above 22,000 were truncated at 22,000, the upper limit of the linear range of the assay.
Time Frame: 2 weeks after the 2nd vaccination (M2.5), 2 weeks after the 3rd vaccination (M6.5), 6 months after the 3rd vaccination (M12)
Population: In this report, the overall number of participants analyzed represents the enrolled participants at 2 weeks after the 2nd vaccination, 2 weeks after the 3rd vaccination, and 6 months after the 3rd vaccination. The Number Analyzed in the Outcome Measure Data Table shows the number of participants with available BAMA data after filtering for assay specific quality control criteria.
Measure: Median (Inter-Quartile Range); unit: Relative fluorescence units
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Relative fluorescence units
  254008_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  254008_D11gp120.avi/293F, 1: 50, M2.5 | 9.75 [1 to 93.5] | 9.5 [1 to 57] | 1 [1 to 30.25] | 65.5 [1 to 491.25] | 173 [1 to 437.25] | 31.38 [5.88 to 494.94]
  254008_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  254008_D11gp120.avi/293F, 1: 50, M6.5 | 133 [10.38 to 489.25] | 418.5 [41.25 to 1273.5] | 105.62 [2.88 to 313.75] | 72.38 [19.38 to 384.88] | 1636 [592 to 2218.5] | 482.75 [279.75 to 2414.75]
  254008_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  254008_D11gp120.avi/293F, 1: 50, M12 | 1 [1 to 3.75] | 1 [1 to 31] | 8.75 [1 to 25.5] | 1 [1 to 1] | 61 [1.63 to 191.12] | 4.5 [1 to 91]
  51802_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  51802_D11gp120.avi/293F, 1: 50, M2.5 | 1 [1 to 19.62] | 1 [1 to 10] | 4.25 [1 to 29.25] | 1 [1 to 1] | 1 [1 to 54] | 8.38 [1 to 70.31]
  51802_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  51802_D11gp120.avi/293F, 1: 50, M6.5 | 1 [1 to 10.31] | 20 [1 to 168.75] | 21.62 [1 to 50.69] | 1 [1 to 1] | 118.75 [2.63 to 375.62] | 99.5 [1 to 314.75]
  51802_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  51802_D11gp120.avi/293F, 1: 50, M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 31.88] | 1 [1 to 1]
  A244 D11gp120_avi, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  A244 D11gp120_avi, 1: 50, M2.5 | 46.5 [6.13 to 292.75] | 10.5 [1 to 131.5] | 11.25 [1 to 190.25] | 19 [1 to 420] | 74.5 [4 to 317.25] | 92.75 [54.25 to 689.81]
  A244 D11gp120_avi, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  A244 D11gp120_avi, 1: 50, M6.5 | 303.62 [129.69 to 696.06] | 180.25 [42.25 to 964.75] | 199 [19.81 to 403.19] | 135 [31.44 to 196.69] | 1482.25 [362.62 to 3138] | 784.5 [237.25 to 2758.25]
  A244 D11gp120_avi, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  A244 D11gp120_avi, 1: 50, M12 | 1 [1 to 6.5] | 10.75 [1 to 78] | 17 [1 to 46.75] | 1 [1 to 60] | 59.75 [6.38 to 144.88] | 33.12 [11.75 to 69.56]
  B.6240_D11gp120/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  B.6240_D11gp120/293F, 1: 50, M2.5 | 8 [1 to 223.62] | 3.5 [1 to 49.25] | 3.75 [1 to 320] | 1 [1 to 33] | 39.5 [1 to 204.5] | 37.25 [1 to 348.94]
  B.6240_D11gp120/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  B.6240_D11gp120/293F, 1: 50, M6.5 | 78.62 [1 to 379.69] | 133.25 [4 to 624.5] | 40.38 [1 to 261.94] | 68.62 [14.94 to 308.44] | 884.5 [328.5 to 2199.5] | 670.5 [167.5 to 2081.25]
  B.6240_D11gp120/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  B.6240_D11gp120/293F, 1: 50, M12 | 1 [1 to 1] | 1 [1 to 12.75] | 1 [1 to 7.75] | 1 [1 to 10] | 13.75 [1 to 166.5] | 1 [1 to 13.94]
  BG505_MD39.3, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3, 1: 50, M2.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [20364.25 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [20303.38 to 22000]
  BG505_MD39.3, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3, 1: 50, M6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [17368.62 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 13 | 15 | 16
  BG505_MD39.3, 1: 50, M12 | 21533.75 [14509.81 to 22000] | 13674.5 [9269.75 to 18157.5] | 18339 [8464.81 to 20661.12] | 22000 [15919.5 to 22000] | 21657 [15333.5 to 22000] | 20110.88 [11982.19 to 21963.25]
  BG505_MD39.3_CD4KO4, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_CD4KO4, 1: 50, M2.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_CD4KO4, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_CD4KO4, 1: 50, M6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [21908.25 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_CD4KO4, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39.3_CD4KO4, 1: 50, M12 | 22000 [22000 to 22000] | 22000 [18783.5 to 22000] | 22000 [17454.88 to 22000] | 22000 [22000 to 22000] | 22000 [21889.25 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M2.5 | 16254.25 [12636.88 to 20457.88] | 11775.5 [9941.25 to 15384] | 12404.5 [11145 to 16712.25] | 15431.75 [10832 to 20131] | 15472.25 [12399.75 to 18047.75] | 15092.38 [9712.5 to 22000]
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M6.5 | 20013.5 [15814.69 to 22000] | 19060.5 [15452 to 22000] | 20087.62 [14704.69 to 22000] | 17648.12 [4395.5 to 22000] | 22000 [21866.5 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M12 | 5045.25 [3281.56 to 7325] | 6951.25 [3752.75 to 8770.25] | 8530.12 [3159.5 to 10593.5] | 5269.75 [4347.94 to 6839.12] | 11112.25 [6684.62 to 13390.88] | 10714.5 [5377.44 to 12897]
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M2.5 | 12200.25 [7355.38 to 15692.88] | 10560.75 [4591.5 to 18965] | 16989.5 [11869 to 20986.75] | 13412.5 [9731.25 to 17226.5] | 22000 [17147.5 to 22000] | 22000 [19720.19 to 22000]
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M6.5 | 21770.38 [18509.38 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 19996 [5802.75 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M12 | 4398 [2621.75 to 5618.25] | 6428.75 [4436 to 14442.5] | 6688.5 [3001 to 15936.75] | 2861.75 [2318 to 4886.25] | 19599.75 [7208.5 to 22000] | 22000 [14025.25 to 22000]
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M2.5 | 16300.75 [11904.88 to 20198.38] | 11121.25 [8643.75 to 15120.75] | 11629 [10107.25 to 15439.75] | 15360.5 [10514.5 to 20268.25] | 13386.5 [11705.25 to 16777.5] | 14496.62 [8994 to 22000]
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M6.5 | 19182.5 [16040.38 to 22000] | 18484.75 [15080 to 22000] | 19112.5 [12667.75 to 22000] | 17901.5 [3917.62 to 22000] | 22000 [21086.38 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 13 | 15 | 16
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M12 | 4491.62 [2907.5 to 6424.19] | 5787.5 [3354.5 to 7598.75] | 7891.62 [2800.38 to 10132.44] | 4480.25 [3464.75 to 5481] | 10265 [6073.62 to 12169.75] | 9672 [4632.19 to 11842.81]
  BG505_MD39.3_pHLsecAvi, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_pHLsecAvi, 1: 50, M2.5 | 9830.75 [5910.12 to 12879.25] | 7920 [4155 to 15617] | 14802.75 [9432.5 to 17777.5] | 10246.5 [7288.75 to 13637] | 21332.25 [14163.5 to 22000] | 22000 [17623.81 to 22000]
  BG505_MD39.3_pHLsecAvi, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_pHLsecAvi, 1: 50, M6.5 | 18019.75 [14887.75 to 20101.12] | 22000 [22000 to 22000] | 22000 [21491.5 to 22000] | 15991.12 [4274.25 to 20183.69] | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  BG505_MD39.3_pHLsecAvi, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BG505_MD39.3_pHLsecAvi, 1: 50, M12 | 3490.5 [2451.75 to 5279.5] | 5952 [4190 to 13786.25] | 6454.75 [2743.75 to 15552] | 2791 [2117.75 to 4520.75] | 19032 [6850.38 to 22000] | 22000 [13301.31 to 22000]
  BG505_MD39_C1-113-125_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 17
  BG505_MD39_C1-113-125_biotin, 1: 50, M2.5 | 275 [108.75 to 481.12] | 162.5 [39.5 to 259.5] | 146.75 [62 to 385.75] | 628 [167.75 to 1148.25] | 291 [65.25 to 929.25] | 185.5 [76.75 to 468.75]
  BG505_MD39_C1-113-125_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39_C1-113-125_biotin, 1: 50, M6.5 | 300.88 [102.94 to 676.62] | 285 [107.5 to 517.5] | 217.62 [96.44 to 952.88] | 896.88 [567.19 to 1525.5] | 507.75 [83.88 to 728.12] | 278.88 [94.19 to 504.81]
  BG505_MD39_C1-113-125_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 15
  BG505_MD39_C1-113-125_biotin, 1: 50, M12 | 232.75 [90 to 543.75] | 175 [71.25 to 388.75] | 275 [110 to 868] | 927.25 [536 to 1675.5] | 286 [83.5 to 733] | 222.5 [122 to 447.38]
  BG505_MD39_HR1-562-577_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 16 | 17
  BG505_MD39_HR1-562-577_biotin, 1: 50, M2.5 | 558.75 [186.62 to 2608.12] | 240.5 [147 to 1160.5] | 207.25 [99.25 to 675.25] | 1836.25 [554.25 to 2746.25] | 557.25 [252.56 to 846.81] | 624.25 [383.25 to 2053.25]
  BG505_MD39_HR1-562-577_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 14 | 16
  BG505_MD39_HR1-562-577_biotin, 1: 50, M6.5 | 488.12 [186.06 to 1544.88] | 466 [224 to 2057.5] | 519.62 [93.75 to 1598.19] | 1430.38 [710.75 to 2019] | 545 [315.56 to 864.94] | 458.62 [333.56 to 2494.38]
  BG505_MD39_HR1-562-577_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 14 | 15
  BG505_MD39_HR1-562-577_biotin, 1: 50, M12 | 385 [254.5 to 1257.75] | 498.5 [192.75 to 1508] | 546.75 [119.25 to 1060.75] | 1213.5 [496.75 to 1655.75] | 395 [215.38 to 881.12] | 698.25 [253 to 1878.38]
  BG505_MD39_HR1-572-587_biotin, 1: 50, M2.5: number analyzed (Participants) | 13 | 16 | 17 | 13 | 17 | 17
  BG505_MD39_HR1-572-587_biotin, 1: 50, M2.5 | 448.5 [158 to 961.75] | 288.38 [156.88 to 759.81] | 351.75 [68.25 to 610] | 893.5 [548.75 to 1389] | 583.25 [207 to 981.5] | 455.25 [220.5 to 1735.75]
  BG505_MD39_HR1-572-587_biotin, 1: 50, M6.5: number analyzed (Participants) | 14 | 16 | 16 | 12 | 15 | 16
  BG505_MD39_HR1-572-587_biotin, 1: 50, M6.5 | 781.62 [206.75 to 1561.75] | 490 [349.69 to 1903.31] | 506.38 [191.12 to 2041.81] | 1372 [774.75 to 1881.81] | 361.5 [135.12 to 1203.75] | 499.12 [171.88 to 4565.44]
  BG505_MD39_HR1-572-587_biotin, 1: 50, M12: number analyzed (Participants) | 15 | 16 | 17 | 13 | 15 | 15
  BG505_MD39_HR1-572-587_biotin, 1: 50, M12 | 191 [144 to 1239.25] | 268.5 [88.5 to 448.56] | 277.25 [113.5 to 882.5] | 1048.25 [531.5 to 1191.75] | 309.25 [101.25 to 709.75] | 330.5 [193 to 1745.25]
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 16 | 13 | 17 | 17
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M2.5 | 215 [151.25 to 621.62] | 160 [57.5 to 237.25] | 175.75 [36.06 to 304.06] | 561 [320 to 1064.75] | 202.5 [46.25 to 501] | 201.5 [80.5 to 522]
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 15 | 12 | 15 | 16
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M6.5 | 254.12 [144 to 1160.06] | 259.75 [88.25 to 488.75] | 134.75 [56.75 to 383.75] | 537.5 [462.44 to 1289.69] | 96.75 [73.62 to 444] | 247.25 [107.88 to 647]
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 16 | 13 | 15 | 15
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M12 | 237.75 [171.25 to 1908] | 236.25 [95 to 543.75] | 273.12 [95.25 to 452] | 847.25 [594.75 to 1293.5] | 249.75 [89.62 to 607.62] | 400.25 [180.38 to 557.38]
  BG505_MD39_V3_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 14 | 17 | 17 | 13 | 17 | 17
  BG505_MD39_V3_peptide_biotin, 1: 50, M2.5 | 13211.12 [5316.88 to 21260.44] | 6695.75 [837 to 10557] | 2331.25 [830.5 to 10837.25] | 11340.75 [5213.25 to 22000] | 15905.75 [6229.75 to 21372.25] | 8418 [2608.5 to 22000]
  BG505_MD39_V3_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 15 | 17 | 16 | 12 | 15 | 16
  BG505_MD39_V3_peptide_biotin, 1: 50, M6.5 | 17530 [8149.88 to 22000] | 22000 [2471 to 22000] | 10530 [4339.31 to 22000] | 13340.5 [2089.19 to 22000] | 22000 [14387.62 to 22000] | 22000 [12141.19 to 22000]
  BG505_MD39_V3_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 15
  BG505_MD39_V3_peptide_biotin, 1: 50, M12 | 2088 [903.12 to 7163.38] | 3303.25 [1742.75 to 8927.25] | 2025.75 [569.5 to 6822.5] | 2612.25 [1977.75 to 4270.25] | 9554 [4095.62 to 12290.5] | 6621.75 [1675.5 to 13496.75]
  BG505_MPER_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MPER_peptide_biotin, 1: 50, M2.5 | 86 [33.5 to 138.5] | 42.75 [11 to 110] | 76.25 [23.25 to 153.5] | 212.5 [85.5 to 312] | 88.25 [31.75 to 136.25] | 66.88 [22.69 to 135.56]
  BG505_MPER_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MPER_peptide_biotin, 1: 50, M6.5 | 140.25 [86.31 to 270.69] | 178.75 [100.25 to 323.75] | 117.62 [68.5 to 249.5] | 339.25 [239.75 to 561.88] | 343.75 [152.38 to 503.88] | 247.5 [186.75 to 428.25]
  BG505_MPER_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BG505_MPER_peptide_biotin, 1: 50, M12 | 47.75 [14.5 to 72] | 20.5 [1 to 131.25] | 50.5 [20 to 114.75] | 233.25 [44 to 436.25] | 87.25 [21.88 to 266.62] | 61 [34.12 to 134.25]
  BJOX002_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BJOX002_D11gp120.avi/293F, 1: 50, M2.5 | 1 [1 to 37.62] | 2 [1 to 15.5] | 1 [1 to 16] | 4.25 [1 to 51.5] | 46.75 [1 to 125.25] | 39.75 [10.69 to 151.38]
  BJOX002_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BJOX002_D11gp120.avi/293F, 1: 50, M6.5 | 109.38 [63 to 206.25] | 154.5 [35.25 to 185.5] | 100.75 [34.94 to 208.25] | 108 [74.12 to 225.19] | 353 [203.38 to 1214.75] | 278 [102.25 to 1425.25]
  BJOX002_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BJOX002_D11gp120.avi/293F, 1: 50, M12 | 1 [1 to 6.75] | 4.5 [1 to 12.75] | 12.75 [1 to 34.25] | 1 [1 to 1] | 6 [1 to 36.12] | 3.63 [1 to 24.5]
  BORI_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BORI_D11gp120.avi/293F, 1: 50, M2.5 | 14.25 [1 to 36.62] | 1 [1 to 4.75] | 1 [1 to 1.5] | 1 [1 to 20.5] | 12.75 [1 to 39.25] | 1 [1 to 26.25]
  BORI_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BORI_D11gp120.avi/293F, 1: 50, M6.5 | 63.88 [21.25 to 72.5] | 49.25 [28 to 126.75] | 50.38 [12.69 to 136.69] | 76.5 [37.12 to 97.5] | 322.75 [121.88 to 781.25] | 169.5 [60 to 565.75]
  BORI_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BORI_D11gp120.avi/293F, 1: 50, M12 | 1 [1 to 39.75] | 2.25 [1 to 25.25] | 16.25 [5.25 to 42.25] | 8.5 [4 to 62] | 34.5 [19.12 to 55] | 19.88 [1 to 41.12]
  CNE20_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  CNE20_D11gp120.avi/293F, 1: 50, M2.5 | 29.75 [1.88 to 90] | 6.5 [1 to 85.75] | 8.5 [1 to 136.25] | 1 [1 to 60.25] | 131.75 [1 to 340.75] | 50 [2.88 to 363]
  CNE20_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  CNE20_D11gp120.avi/293F, 1: 50, M6.5 | 104.5 [1 to 300.94] | 244.75 [13.25 to 683.75] | 164.25 [1 to 337.62] | 46.75 [17.62 to 249.12] | 1164 [447.62 to 1986.75] | 450 [138 to 2473.5]
  CNE20_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  CNE20_D11gp120.avi/293F, 1: 50, M12 | 1 [1 to 1] | 1 [1 to 7] | 8.25 [1 to 41.25] | 1 [1 to 46] | 43.5 [1.88 to 129.25] | 1 [1 to 77.81]
  Link14_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 17
  Link14_peptide_biotin, 1: 50, M2.5 | 1213 [361.38 to 1924] | 179.25 [55.75 to 450.75] | 165.25 [33.25 to 365.5] | 1727.5 [1115.5 to 3608.25] | 389.25 [112.5 to 539.25] | 223.5 [83.25 to 440.5]
  Link14_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  Link14_peptide_biotin, 1: 50, M6.5 | 792.25 [573.75 to 2124.38] | 309.5 [108.25 to 1008.75] | 212.62 [89.81 to 453.62] | 1896.12 [1012.12 to 2339.56] | 488.75 [154.38 to 818.5] | 281.88 [94.06 to 499.88]
  Link14_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 15
  Link14_peptide_biotin, 1: 50, M12 | 222.25 [95 to 977.75] | 113.75 [68.75 to 406.25] | 136.25 [86.5 to 414] | 1258.5 [498 to 1556] | 182 [101.25 to 423.62] | 189.75 [103.88 to 358.12]
  TT31P.2792_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  TT31P.2792_D11gp120.avi/293F, 1: 50, M2.5 | 1 [1 to 65.38] | 1 [1 to 38.5] | 1 [1 to 159.75] | 13.25 [1 to 147.25] | 35.5 [1 to 356.25] | 50.62 [6.06 to 431.56]
  TT31P.2792_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  TT31P.2792_D11gp120.avi/293F, 1: 50, M6.5 | 60.75 [1 to 887.5] | 259.75 [10.5 to 484] | 121 [1 to 534.19] | 48.88 [26.44 to 343.62] | 1527.75 [504.75 to 2062.38] | 917.75 [226.5 to 1802.75]
  TT31P.2792_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  TT31P.2792_D11gp120.avi/293F, 1: 50, M12 | 1 [1 to 1] | 2 [1 to 29.75] | 8 [1 to 32.25] | 1 [1 to 1] | 37.5 [1.38 to 75.38] | 8.63 [1 to 58.25]
  gp41, 1: 50, M2.5: number analyzed (Participants) | 14 | 17 | 16 | 13 | 17 | 18
  gp41, 1: 50, M2.5 | 619.12 [400.12 to 1077.06] | 435.75 [165.75 to 1014.5] | 400.62 [132 to 791] | 1374.25 [656.5 to 1881.25] | 749.25 [449.75 to 1086.5] | 786.88 [532 to 1475]
  gp41, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 14 | 12 | 14 | 17
  gp41, 1: 50, M6.5 | 989 [748.38 to 2367.56] | 1578.75 [904 to 1666.75] | 1455 [658.94 to 2155] | 2305.25 [1630.5 to 4427.44] | 1421.12 [822.19 to 2716.62] | 1348.25 [939.25 to 2433.75]
  gp41, 1: 50, M12: number analyzed (Participants) | 15 | 17 | 15 | 12 | 15 | 15
  gp41, 1: 50, M12 | 1020.25 [862.75 to 2139.5] | 1378.5 [895.25 to 1755.5] | 1016.5 [734.5 to 1308.12] | 2721.75 [1422.62 to 3349.75] | 907.5 [635.25 to 1945.25] | 1713.75 [861.38 to 2506.12]
  scrambled_MD39_peptide-biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 15 | 17
  scrambled_MD39_peptide-biotin, 1: 50, M2.5 | 184 [140.5 to 1433.25] | 229 [59 to 630] | 277.5 [145.5 to 417.75] | 593.5 [329.75 to 1083.5] | 549.75 [71.5 to 794.62] | 454.5 [94.75 to 843.75]
  scrambled_MD39_peptide-biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 13 | 16
  scrambled_MD39_peptide-biotin, 1: 50, M6.5 | 245.12 [152.5 to 1823.62] | 346.25 [194.75 to 795.25] | 423.38 [287.69 to 1141.25] | 863.62 [484.81 to 1769.25] | 538.5 [103.75 to 762] | 477.5 [95.25 to 1049.12]
  scrambled_MD39_peptide-biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 13 | 15
  scrambled_MD39_peptide-biotin, 1: 50, M12 | 255.5 [156 to 1484.25] | 398.75 [250 to 942.75] | 522.75 [220 to 1130.75] | 720 [548.25 to 1680.5] | 709.75 [174.5 to 981] | 437.5 [198 to 936]

22. Secondary Outcome: Response Rate Serum IgG Binding Antibodies to the BG505 Trimer, and Specific Epitopes (Base of Trimer, V3, Internal Epitope) as Measured by Binding Antibody Multiplex Assay (BAMA)
Description: as for outcome 21
Time Frame: as for outcome 21
Population: In this report, the overall number of participants analyzed represents the enrolled participants at 2 weeks after the 2nd vaccination, 2 weeks after the 3rd vaccination and 6 months after the 3rd vaccination. The Number Analyzed in the Outcome Measure Data Table shows the number of participants with available BAMA data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  254008_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  254008_D11gp120.avi/293F, 1: 50, M2.5 | 3 | 4 | 2 | 6 | 9 | 8
  254008_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  254008_D11gp120.avi/293F, 1: 50, M6.5 | 8 | 11 | 8 | 5 | 12 | 14
  254008_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  254008_D11gp120.avi/293F, 1: 50, M12 | 2 | 3 | 2 | 2 | 5 | 4
  51802_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  51802_D11gp120.avi/293F, 1: 50, M2.5 | 2 | 0 | 1 | 1 | 2 | 4
  51802_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  51802_D11gp120.avi/293F, 1: 50, M6.5 | 1 | 7 | 1 | 0 | 9 | 8
  51802_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  51802_D11gp120.avi/293F, 1: 50, M12 | 1 | 1 | 0 | 0 | 1 | 1
  A244 D11gp120_avi, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  A244 D11gp120_avi, 1: 50, M2.5 | 4 | 5 | 3 | 4 | 7 | 8
  A244 D11gp120_avi, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  A244 D11gp120_avi, 1: 50, M6.5 | 11 | 11 | 10 | 7 | 12 | 16
  A244 D11gp120_avi, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  A244 D11gp120_avi, 1: 50, M12 | 3 | 2 | 3 | 1 | 4 | 3
  B.6240_D11gp120/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  B.6240_D11gp120/293F, 1: 50, M2.5 | 3 | 2 | 2 | 2 | 3 | 5
  B.6240_D11gp120/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  B.6240_D11gp120/293F, 1: 50, M6.5 | 5 | 8 | 6 | 4 | 11 | 12
  B.6240_D11gp120/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  B.6240_D11gp120/293F, 1: 50, M12 | 1 | 2 | 0 | 1 | 4 | 1
  BG505_MD39.3, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3, 1: 50, M2.5 | 15 | 15 | 16 | 13 | 17 | 16
  BG505_MD39.3, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3, 1: 50, M6.5 | 16 | 16 | 16 | 11 | 15 | 16
  BG505_MD39.3, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 13 | 15 | 16
  BG505_MD39.3, 1: 50, M12 | 16 | 16 | 16 | 12 | 15 | 15
  BG505_MD39.3_CD4KO4, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_CD4KO4, 1: 50, M2.5 | 15 | 15 | 16 | 13 | 17 | 16
  BG505_MD39.3_CD4KO4, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_CD4KO4, 1: 50, M6.5 | 16 | 16 | 16 | 11 | 15 | 16
  BG505_MD39.3_CD4KO4, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39.3_CD4KO4, 1: 50, M12 | 16 | 16 | 16 | 12 | 15 | 16
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M2.5 | 14 | 15 | 16 | 10 | 17 | 16
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M6.5 | 16 | 16 | 16 | 10 | 15 | 16
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39.3_CD4KO4_baseKO_1CCv4, 1: 50, M12 | 16 | 16 | 15 | 11 | 15 | 15
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M2.5 | 15 | 16 | 17 | 12 | 17 | 16
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M6.5 | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BG505_MD39.3_CD4KO4_pHLsecAvi, 1: 50, M12 | 17 | 17 | 17 | 12 | 15 | 15
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M2.5 | 14 | 15 | 16 | 10 | 17 | 16
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M6.5 | 16 | 16 | 16 | 10 | 15 | 16
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 16 | 13 | 15 | 16
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M12 | 15 | 16 | 15 | 11 | 15 | 15
  BG505_MD39.3_pHLsecAvi, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MD39.3_pHLsecAvi, 1: 50, M2.5 | 15 | 16 | 17 | 12 | 17 | 16
  BG505_MD39.3_pHLsecAvi, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MD39.3_pHLsecAvi, 1: 50, M6.5 | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39.3_pHLsecAvi, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BG505_MD39.3_pHLsecAvi, 1: 50, M12 | 17 | 17 | 17 | 12 | 15 | 15
  BG505_MD39_C1-113-125_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 17
  BG505_MD39_C1-113-125_biotin, 1: 50, M2.5 | 0 | 0 | 0 | 0 | 0 | 0
  BG505_MD39_C1-113-125_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  BG505_MD39_C1-113-125_biotin, 1: 50, M6.5 | 0 | 0 | 1 | 0 | 0 | 0
  BG505_MD39_C1-113-125_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 15
  BG505_MD39_C1-113-125_biotin, 1: 50, M12 | 0 | 0 | 2 | 2 | 0 | 0
  BG505_MD39_HR1-562-577_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 16 | 17
  BG505_MD39_HR1-562-577_biotin, 1: 50, M2.5 | 3 | 0 | 1 | 1 | 1 | 0
  BG505_MD39_HR1-562-577_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 14 | 16
  BG505_MD39_HR1-562-577_biotin, 1: 50, M6.5 | 2 | 1 | 1 | 0 | 1 | 0
  BG505_MD39_HR1-562-577_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 14 | 15
  BG505_MD39_HR1-562-577_biotin, 1: 50, M12 | 0 | 1 | 3 | 1 | 0 | 1
  BG505_MD39_HR1-572-587_biotin, 1: 50, M2.5: number analyzed (Participants) | 13 | 16 | 17 | 13 | 17 | 17
  BG505_MD39_HR1-572-587_biotin, 1: 50, M2.5 | 0 | 0 | 1 | 0 | 0 | 1
  BG505_MD39_HR1-572-587_biotin, 1: 50, M6.5: number analyzed (Participants) | 14 | 16 | 16 | 12 | 15 | 16
  BG505_MD39_HR1-572-587_biotin, 1: 50, M6.5 | 0 | 0 | 2 | 0 | 0 | 1
  BG505_MD39_HR1-572-587_biotin, 1: 50, M12: number analyzed (Participants) | 15 | 16 | 17 | 13 | 15 | 15
  BG505_MD39_HR1-572-587_biotin, 1: 50, M12 | 0 | 0 | 1 | 1 | 0 | 1
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 16 | 13 | 17 | 17
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M2.5 | 0 | 0 | 0 | 0 | 0 | 0
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 15 | 12 | 15 | 16
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M6.5 | 0 | 0 | 0 | 0 | 0 | 0
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 16 | 13 | 15 | 15
  BG505_MD39_HR1-582-597_peptide_biotin, 1: 50, M12 | 0 | 1 | 1 | 1 | 0 | 0
  BG505_MD39_V3_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 14 | 17 | 17 | 13 | 17 | 17
  BG505_MD39_V3_peptide_biotin, 1: 50, M2.5 | 11 | 8 | 7 | 10 | 14 | 11
  BG505_MD39_V3_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 15 | 17 | 16 | 12 | 15 | 16
  BG505_MD39_V3_peptide_biotin, 1: 50, M6.5 | 13 | 12 | 13 | 8 | 13 | 14
  BG505_MD39_V3_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 16 | 17 | 17 | 13 | 15 | 15
  BG505_MD39_V3_peptide_biotin, 1: 50, M12 | 4 | 8 | 6 | 6 | 10 | 10
  BG505_MPER_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BG505_MPER_peptide_biotin, 1: 50, M2.5 | 0 | 0 | 0 | 0 | 0 | 0
  BG505_MPER_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BG505_MPER_peptide_biotin, 1: 50, M6.5 | 1 | 0 | 0 | 0 | 0 | 0
  BG505_MPER_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BG505_MPER_peptide_biotin, 1: 50, M12 | 0 | 0 | 1 | 1 | 0 | 0
  BJOX002_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BJOX002_D11gp120.avi/293F, 1: 50, M2.5 | 1 | 2 | 2 | 2 | 6 | 6
  BJOX002_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BJOX002_D11gp120.avi/293F, 1: 50, M6.5 | 8 | 10 | 8 | 6 | 13 | 13
  BJOX002_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BJOX002_D11gp120.avi/293F, 1: 50, M12 | 1 | 0 | 0 | 1 | 2 | 2
  BORI_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  BORI_D11gp120.avi/293F, 1: 50, M2.5 | 1 | 0 | 2 | 2 | 2 | 4
  BORI_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  BORI_D11gp120.avi/293F, 1: 50, M6.5 | 2 | 6 | 5 | 2 | 11 | 10
  BORI_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  BORI_D11gp120.avi/293F, 1: 50, M12 | 1 | 1 | 0 | 0 | 1 | 2
  CNE20_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  CNE20_D11gp120.avi/293F, 1: 50, M2.5 | 3 | 4 | 2 | 2 | 8 | 7
  CNE20_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  CNE20_D11gp120.avi/293F, 1: 50, M6.5 | 7 | 10 | 8 | 4 | 13 | 14
  CNE20_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  CNE20_D11gp120.avi/293F, 1: 50, M12 | 1 | 2 | 1 | 1 | 5 | 3
  Link14_peptide_biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 17
  Link14_peptide_biotin, 1: 50, M2.5 | 1 | 0 | 0 | 4 | 0 | 0
  Link14_peptide_biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 16
  Link14_peptide_biotin, 1: 50, M6.5 | 2 | 2 | 0 | 2 | 0 | 0
  Link14_peptide_biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 15
  Link14_peptide_biotin, 1: 50, M12 | 1 | 0 | 1 | 1 | 0 | 0
  TT31P.2792_D11gp120.avi/293F, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 17 | 18
  TT31P.2792_D11gp120.avi/293F, 1: 50, M2.5 | 2 | 1 | 4 | 4 | 8 | 7
  TT31P.2792_D11gp120.avi/293F, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 15 | 17
  TT31P.2792_D11gp120.avi/293F, 1: 50, M6.5 | 5 | 10 | 8 | 3 | 12 | 15
  TT31P.2792_D11gp120.avi/293F, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 15 | 16
  TT31P.2792_D11gp120.avi/293F, 1: 50, M12 | 2 | 1 | 1 | 1 | 2 | 3
  gp41, 1: 50, M2.5: number analyzed (Participants) | 14 | 17 | 16 | 13 | 17 | 18
  gp41, 1: 50, M2.5 | 1 | 0 | 0 | 0 | 0 | 1
  gp41, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 14 | 12 | 14 | 17
  gp41, 1: 50, M6.5 | 3 | 2 | 2 | 2 | 2 | 3
  gp41, 1: 50, M12: number analyzed (Participants) | 15 | 17 | 15 | 12 | 15 | 15
  gp41, 1: 50, M12 | 1 | 3 | 0 | 1 | 1 | 2
  scrambled_MD39_peptide-biotin, 1: 50, M2.5: number analyzed (Participants) | 15 | 17 | 17 | 13 | 15 | 17
  scrambled_MD39_peptide-biotin, 1: 50, M2.5 | 0 | 0 | 0 | 0 | 0 | 0
  scrambled_MD39_peptide-biotin, 1: 50, M6.5: number analyzed (Participants) | 16 | 17 | 16 | 12 | 13 | 16
  scrambled_MD39_peptide-biotin, 1: 50, M6.5 | 0 | 0 | 0 | 0 | 0 | 0
  scrambled_MD39_peptide-biotin, 1: 50, M12: number analyzed (Participants) | 17 | 17 | 17 | 13 | 13 | 15
  scrambled_MD39_peptide-biotin, 1: 50, M12 | 0 | 1 | 1 | 1 | 0 | 0

23. Secondary Outcome: Magnitude of CD4+ T-cell Responses as Assessed by Intracellular Cytokine Staining Assays (ICS)
Description: Flow cytometry was used to examine HIV-1-specific CD4+ T-cell responses using a validated the 27-color COVID v2 staining panel. Response magnitudes were defined as the negative control- or background adjusted percent of CD4+ T cells expressing the cytokines or cytokine combinations. Total Env is the sum of gp120 and gp41 peptide pools. One-sided Fisher's exact test was applied to test whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. A multiplicity adjustment was made to the individual peptide pool p-values using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was ≤ 0.00001, the response to the peptide pool for the T-cell subset was considered positive. Records are excluded if the number of CD4+ T-cell subsets is less than ten thousands
Time Frame: 2 weeks after the 3rd vaccination (M6.5)
Population: In this report, the overall number of participants analyzed represents the enrolled participants at 2 weeks after the 3rd vaccination. The Number Analyzed in the Outcome Measure Data Table shows the number of participants with available ICS data after filtering for assay specific quality control criteria.
Measure: Median (Inter-Quartile Range); unit: Percent T-cells expressing cytokines
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Percent T-cells expressing cytokines
  BG505 MD39.3 gp120, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp120, IFN-γ and/or IL-2, M6.5 | 0.2 [0.1 to 0.3] | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.5] | 0.1 [0.1 to 0.3] | 0.3 [0.3 to 0.4] | 0.3 [0.1 to 0.6]
  BG505 MD39.3 gp120, IL-21, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp120, IL-21, M6.5 | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0.1] | 0 [0 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0 to 0.1]
  BG505 MD39.3 gp120, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp120, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  BG505 MD39.3 gp41, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp41, IFN-γ and/or IL-2, M6.5 | 0.1 [0 to 0.1] | 0.1 [0 to 0.2] | 0.1 [0 to 0.1] | 0 [0 to 0] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.2]
  BG505 MD39.3 gp41, IL-21, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp41, IL-21, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  BG505 MD39.3 gp41, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp41, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  BG505-MD39.3 gp140 protein, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  BG505-MD39.3 gp140 protein, IFN-γ and/or IL-2, M6.5 | 0.2 [0.1 to 0.2] | 0.1 [0 to 0.1] | 0.2 [0.2 to 0.3] | 0.1 [0.1 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  BG505-MD39.3 gp140 protein, IL-21, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  BG505-MD39.3 gp140 protein, IL-21, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  BG505-MD39.3 gp140 protein, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  BG505-MD39.3 gp140 protein, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  LeadSeq mRNA, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  LeadSeq mRNA, IFN-γ and/or IL-2, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  LeadSeq mRNA, IL-21, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  LeadSeq mRNA, IL-21, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  LeadSeq mRNA, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  LeadSeq mRNA, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Total Env, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  Total Env, IFN-γ and/or IL-2, M6.5 | 0.2 [0.1 to 0.4] | 0.3 [0.2 to 0.4] | 0.3 [0.2 to 0.6] | 0.2 [0.1 to 0.4] | 0.4 [0.3 to 0.5] | 0.5 [0.2 to 0.7]
  Total Env, IL-21, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  Total Env, IL-21, M6.5 | 0 [0 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2]
  Total Env, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  Total Env, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 0 [0 to 0] | 0 [0 to 0.1] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0.1] | 0 [0 to 0.1]

24. Secondary Outcome: Response Rate of CD4+ T-cell Responses as Assessed by Intracellular Cytokine Staining Assays (ICS)
Description: as for outcome 23
Time Frame: 2 weeks after the 3rd vaccination (M6.5)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
Number analyzed (Participants) | 18 | 19 | 17 | 18 | 18 | 18
Participants
  BG505 MD39.3 gp120, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp120, IFN-γ and/or IL-2, M6.5 | 12 | 16 | 14 | 10 | 14 | 16
  BG505 MD39.3 gp120, IL-21, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp120, IL-21, M6.5 | 10 | 12 | 10 | 6 | 11 | 14
  BG505 MD39.3 gp120, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp120, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 6 | 11 | 9 | 5 | 10 | 10
  BG505 MD39.3 gp41, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp41, IFN-γ and/or IL-2, M6.5 | 11 | 14 | 13 | 5 | 12 | 14
  BG505 MD39.3 gp41, IL-21, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp41, IL-21, M6.5 | 3 | 2 | 1 | 1 | 3 | 9
  BG505 MD39.3 gp41, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  BG505 MD39.3 gp41, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 1 | 7 | 2 | 0 | 5 | 3
  BG505-MD39.3 gp140 protein, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  BG505-MD39.3 gp140 protein, IFN-γ and/or IL-2, M6.5 | 4 | 5 | 4 | 4 | 8 | 7
  BG505-MD39.3 gp140 protein, IL-21, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  BG505-MD39.3 gp140 protein, IL-21, M6.5 | 4 | 0 | 2 | 2 | 3 | 4
  BG505-MD39.3 gp140 protein, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  BG505-MD39.3 gp140 protein, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 3 | 3 | 1 | 1 | 4 | 4
  LeadSeq mRNA, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  LeadSeq mRNA, IFN-γ and/or IL-2, M6.5 | 0 | 0 | 0 | 0 | 0 | 0
  LeadSeq mRNA, IL-21, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  LeadSeq mRNA, IL-21, M6.5 | 0 | 0 | 0 | 0 | 0 | 0
  LeadSeq mRNA, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 5 | 7 | 4 | 5 | 8 | 8
  LeadSeq mRNA, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 0 | 0 | 0 | 0 | 0 | 0
  Total Env, IFN-γ and/or IL-2, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  Total Env, IFN-γ and/or IL-2, M6.5 | 12 | 16 | 14 | 10 | 14 | 16
  Total Env, IL-21, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  Total Env, IL-21, M6.5 | 10 | 12 | 10 | 7 | 11 | 14
  Total Env, IL-4 or IL-5 or IL-13 and CD154, M6.5: number analyzed (Participants) | 15 | 17 | 15 | 12 | 14 | 17
  Total Env, IL-4 or IL-5 or IL-13 and CD154, M6.5 | 6 | 11 | 9 | 5 | 10 | 10

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected over a period of 30 days after each vaccination. The Solicited AE assessment were collected through 7 full days after each vaccination. A limited set of AEs, including SAEs, were collected and reported through the end of the main study (Month 12).
Arm/Group | Part A, Group 1: Treatment | Part A, Group 2: Treatment | Part A, Group 3: Treatment | Part B, Group 4: Treatment | Part B, Group 5: Treatment | Part B, Group 6: Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/17 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/19 | 1/17 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 18/18 | 19/19 | 17/17 | 18/18 | 18/18 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: Treatment (N=18) | Part A, Group 2: Treatment (N=19) | Part A, Group 3: Treatment (N=17) | Part B, Group 4: Treatment (N=18) | Part B, Group 5: Treatment (N=18) | Part B, Group 6: Treatment (N=18)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: Treatment (N=18) | Part A, Group 2: Treatment (N=19) | Part A, Group 3: Treatment (N=17) | Part B, Group 4: Treatment (N=18) | Part B, Group 5: Treatment (N=18) | Part B, Group 6: Treatment (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inner ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Solicited) (Gastrointestinal disorders) | 4 (7) | 3 (6) | 8 (13) | 7 (10) | 9 (14) | 10 (16)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chills (Solicited) (General disorders) | 11 (16) | 6 (11) | 11 (17) | 7 (9) | 16 (23) | 13 (17)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (Solicited) (General disorders) | 16 (34) | 12 (26) | 15 (38) | 15 (29) | 18 (40) | 15 (31)
Injection site erythema (Solicited) (General disorders) | 1 (1) | 6 (10) | 1 (2) | 2 (2) | 3 (3) | 6 (8)
Injection site pain (Solicited) (General disorders) | 18 (49) | 18 (47) | 16 (46) | 18 (37) | 18 (49) | 18 (49)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (Solicited) (General disorders) | 2 (3) | 4 (5) | 5 (9) | 4 (4) | 1 (3) | 4 (6)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spirochaetal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Body temperature increased (Solicited) (Investigations) | 4 (4) | 6 (8) | 0 (0) | 1 (2) | 6 (8) | 9 (13)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 8 (13) | 9 (12) | 12 (18) | 7 (10) | 10 (13) | 11 (16)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 13 (22) | 8 (15) | 12 (23) | 11 (18) | 18 (34) | 18 (31)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Solicited) (Nervous system disorders) | 14 (21) | 13 (27) | 14 (29) | 15 (26) | 17 (33) | 17 (32)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Substance use disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine malposition (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT05217641/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT05217641/SAP_001.pdf